CLINICAL TRIAL: NCT05076682
Title: Reverse Triple Negative Immune Resistant Breast Cancer
Acronym: Renaissance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2107239-9
Record Dates: First submitted 2021-09-12; First posted 2021-10-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Triple-negative Breast Cancer
Keywords: TNBC; molecular subtype; precision Treatment; immunotherapy; choline; sodium cromoglicate; efavirenz
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Choline; Drug Therapy; Cromolyn Sodium; efavirenz; pegylated granulocyte colony-stimulating factor; Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Choline (Experimental): Choline with anti-PD-1 immunotherapy
  Interventions: Drug: Choline; Drug: anti-PD-1 antibody and chemotherapy
- Sodium cromoglicate (Experimental): Sodium cromoglicate with anti-PD-1 immunotherapy
  Interventions: Drug: anti-PD-1 antibody and chemotherapy; Drug: Sodium Cromoglicate
- Efavirenz (Experimental): Efavirenz with anti-PD-1 immunotherapy
  Interventions: Drug: anti-PD-1 antibody and chemotherapy; Drug: Efavirenz
- HER2 low (Experimental): HER2 low expression
  Interventions: Drug: SHR-A1811; Drug: SHR-1316
- HER2 0 (Experimental): HER2 0 expression
  Interventions: Drug: SHR-A2102; Drug: SHR-1316
- AK131 (Experimental): AK131(CD73/PD1 bispecific antibody)
  Interventions: Drug: AK131
- Mecapegfilgrastim (Experimental): Mecapegfilgrastim with anti-PD-1 immunotherapy
  Interventions: Drug: anti-PD-1 antibody and chemotherapy; Drug: Mecapegfilgrastim
- Theophylline (Experimental): Theophylline with anti-PD-1 immunotherapy
  Interventions: Drug: Theophylline

INTERVENTIONS:
Drug: Choline — Choline 300mg tid or 500mg bid, p.o
  Arms: Choline
Drug: anti-PD-1 antibody and chemotherapy — PD-1 antibody SHR1210 200mg q2w chemotherapy (whether and which should be given depends on the treatment regimen before enrollment)
  Arms: Choline; Efavirenz; Mecapegfilgrastim; Sodium cromoglicate
Drug: Sodium Cromoglicate — Sodium Cromoglicate will be administered intranasally (nasal spray) (5 spray each nostril 4 times a day, 1 mg/spray)
  Arms: Sodium cromoglicate
Drug: Efavirenz — Efavirenz 600mg qd, p.o
  Arms: Efavirenz
Drug: SHR-A1811 — 4.8mg/kg q3w
  Arms: HER2 low
Drug: SHR-A2102 — 6mg/kg q3w
  Arms: HER2 0
Drug: SHR-1316 — 1200mg q3w
  Arms: HER2 0; HER2 low
Drug: Mecapegfilgrastim — Mecapegfilgrastim, 6mg, d3, q3w, s.c.
  Arms: Mecapegfilgrastim
Drug: AK131 — AK131, 40mg/kg i.v., q2w
  Arms: AK131
Drug: Theophylline — Theophylline, 100mg bid, p.o.
  Arms: Theophylline

SUMMARY:
This is a Phase II, open-label, seven-arm parallel study evaluating the efficacy and safety of combined treatment (sodium cromoglicate, choline, efavirenz, SHR 1811, SHR 2102, mecapegfilgrastim, theophylline) with immune checkpoint inhibitor or immune checkpoint inhibitor rechallenge(AK131) in mTNBC (triple negative breast cancer) patients who progressed during previous immune checkpoint inhibitors.

DETAILED DESCRIPTION:
This is a Phase II, open-label, three-arm parallel study evaluating the efficacy and safety of combined treatment (sodium cromoglicate, choline, efavirenz, SHR 1811, SHR 2102, mecapegfilgrastim) with immune checkpoint inhibitor or immune checkpoint inhibitor rechallenge(AK131) in mTNBC (triple negative breast cancer) patients who progressed during or following previous immune checkpoint inhibitors. The investigators have achieved a breakthrough in the FUTURE study with an ORR (objective response rate) reaching 52.6% in IM (immunomodulatory) subtype TNBC patients. Despite this, there are still some IM subtype patients resistant to immunotherapy. How to reverse immunotherapy resistance or how to increase the sensitivity of immunotherapy efficacy, has become an urgent clinical problem to be solved. The preclinical results of our center show that sodium cromoglicate, choline, efavirenz, SHR 1811, SHR 2102, mecapegfilgrastim, AK131, theophylline play a potentially important role in regulating the tumor immune microenvironment and can inhibit the growth of tumors in mice, and enhance the efficacy of PD-1 inhibitors in mice. Based on preclinical studies, the investigators designed this study to enroll mTNBC patients who have progressed during or following immunotherapy, and to explore the efficacy of these drugs at a clinical level, providing new strategies of combined treatment for TNBC patients.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0, 1, or 2
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Radiologic/objective evidence of recurrence or disease progression after immunotherapy(combined with targeted therapy or chemo ) for metastatic breast cancer(MBC)
* Adequate hematologic and end-organ function, laboratory test results, obtained within 14 days prior to initiation of study treatment.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
* have the cognitive ability to understand the protocol and be willing to participate and to be followed up.

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing CNS metastases
* Active or history of autoimmune disease or immune deficiency
* Significant cardiovascular disease
* History of malignancy other than breast cancer within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Treatment with chemotherapy, radiotherapy,immunotherapy or surgery (outpatient clinic surgery excluded) within 3 weeks prior to initiation of study treatment.
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* History of allergies to the drug components of this trial
* History of eosinophilosis or mastocytosis
* Patients who have been using oral steroid hormones for a long time will need to stop for 4 weeks if they have used them occasionally in the past
* For the Mecapegfilgrastim group, patients had previously received PEG-rhG-CSF in combination with immunotherapy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
Immune changes in peripheral blood | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Baseline through end of study, assessed up to 6 months
Progression Free Survival (PFS) | Randomization to death from any cause, through the end of study,assessed up to 6 months
Safety and treatment-related AEs | Randomization to death from any cause, through the end of study,assessed up to 12 months
Biomarker analysis1 | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Mast cell function will be measured in pretreatment tissues to predict therapy response.
Biomarker analysis2 | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Immunohistochemical staining of pre- and post-treatment tissue sections was carried out to evaluate PD-L1 expression, mast cell function, innate lymphoid cell porprotion and activity, and overall inflammatory status
Biomarker analysis3 | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  The quantity and function of innate lympoid cells will be measured in tissues and/or peripheral blood before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Professor, Principal Investigator — Fudan U
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Wu SY, Jin X, Liu Y, Wang ZY, Zuo WJ, Ma D, Xiao Y, Fu T, Xiao YL, Chen L, Liu XY, Fan L, Wang ZH, Shen M, Liu R, Chai WJ, Shao ZM, Jiang YZ. Mobilizing antigen-presenting mast cells in anti-PD-1-refractory triple-negative breast cancer: a phase 2 trial. Nat Med. 2025 Jul;31(7):2405-2415. doi: 10.1038/s41591-025-03776-7. Epub 2025 Jun 25. PMID 40563015